CLINICAL TRIAL: NCT06615791
Title: FIT FIRST Teen Effectiveness and School Implementation Study - a Cluster Randomised Mixed Methods Trial.
Brief Title: FIT FIRST Teen - School Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other); Team Denmark (Other); The Danish Sports Confederation (Unknown)
Responsible Party: Principal Investigator, Peter Krustrup, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USouthernDenmark-FITFIRSTTeen
Record Dates: First submitted 2024-09-13; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Primary Prevention
Keywords: physical activity; sports
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIT FIRST Teen (Experimental): School teachers will attend a one-day training course and will be given the FIT FIRST Teen manual, which will contain all the activities to be provided during physical education.
  Three 45-minute lessons per week for an entire school year will be administered to students by their teachers.
  Interventions: Behavioral: FIT FIRST Teen
- Control (No Intervention): School teachers will continue to offer the usual physical education curricula to students.

INTERVENTIONS:
Behavioral: FIT FIRST Teen — High intensity sports drills and games.
  Arms: FIT FIRST Teen

SUMMARY:
The goal of this cluster randomised controlled trial is to investigate the effects of the FIT FIRST Teen program on adolescents' physical fitness, motivation, and well-being, as well as the implementation of such a program within schools. The main questions it aims to answer are:

Research Question 1: Does the FIT FIRST Teen program improve cardiorespiratory fitness, body composition, and muscle strength among adolescents?

Research Question 2: Does the FIT FIRST Teen program improve well-being, motivation towards physical activity, and body image among adolescents?

Research Question 3: What are the challenges that teachers and schools will face regarding the implementation of the FIT FIRST Teen program?

The research team will compare the FIT FIRST Teen program to a control (usual physical education curricula) to see if such a program improves adolescents' physical fitness, motivation, and well-being. Participating schools will:

* Participate in a training course, where the core principles of the FIT FIRST Teen program will be delivered.
* Implement the FIT FIRST Teen program for a full school year (three 45-minute lessons a week).
* Keep a logbook where the weekly practised activities will be reported.

DETAILED DESCRIPTION:
Background. Physical activity (PA) is an important part of a healthy lifestyle for children and youth, as it improves physical fitness, motor competencies, and well-being, and reduces the risk of developing overweight and non-communicable diseases later in life. Current recommendations from the Danish Health Authorities are that young people should participate in at least 60 minutes of moderate-to-vigorous physical activity (MVPA) per day, of which at least 3 times per week should involve muscle strengthening training, however, currently only about one-quarter of the Danish 11-15-year-olds meet these recommendations.

Given that children and adolescents, irrespective of socio-economic background, spend a substantial portion of their waking hours in school, schools serve as pivotal settings for the widespread promotion of PA. However, current school-based PA interventions have shown limited effects. Often the poor results of interventions can be ascribed to implementation challenges, encompassing deficiencies in program fidelity, suboptimal attendance rates, or lack of access to intended resources, time, or space. Details about the contextual environment and how to implement interventions are typically derived from implementation evaluations. Nonetheless, such evaluations are rarely undertaken.

The FIT FIRST program was developed to address these limitations. FIT FIRST was originally an acronym for a 40-week intervention study for 8- to 9-year-olds with Frequent Intense Training through Football, Interval Running, and Circuit Strength Training. In 2018, the FIT FIRST 10 concept was developed for 6-9-yr-olds that covered 10 sports. In 2020, the FIT FIRST 20 concept for 10-12-year-olds was developed to include 20 sports. In brief, all versions of the FIT FIRST concept are built on the principles of using multiple sporting activities modified for the school setting, with a focus on high intensity, high involvement, fun, and inclusion. The use of multiple sporting activities modified for the school setting may also recess activities and leisure-time sports. Therefore, it will be investigated whether the developed abilities and motivation for FIT FIRST sporting activities can result in recruitment or re-recruitment of members to the local sports clubs.

The implementation of the FIT FIRST Teen project is based on training teachers to deliver such a program, which has been developed by experienced staff from SDU (University of Southern Denmark (SDU), The DIF (Danish Sports Confederation (DIF), and Team Denmark. These partners have developed 3-6 lessons for each of the sports, all using pair-based exercises and small-sided game drills and activities. All the lessons included in the FIT FIRST Teen program have been developed to (1) provide high-intensity strength and cardiovascular training and (2) motivate children to participate, according to the self-determination theory.

FIT FIRST Teen will run over a full school year with physical fitness, motivation, and well-being as primary outcomes, and project implementation as co-primary outcome. In this study, the research team will be testing the effects of the FIT FIRST Teen program by randomizing schools into two groups. Hence, this will be a cluster RCT with a 1:1 randomization of schools into an intervention arm, which will implement the FIT FIRST Teen program 3 times a week weekly (three 40-minute lessons a week), and a control arm, which will provide the usual physical education curricula.

Measures. To evaluate the intervention effect on adolescents' fitness levels and health profile the following measures will be employed.

Cardiometabolic fitness. The Yo-Yo intermittent recovery level 1 test for adolescents (YYIR1C test) will be conducted to evaluate cardiometabolic fitness levels. Resting heart rate and blood pressure will be measured at rest. We will conduct 3 measurements after an 8-minute resting period.

Body Composition: Tanita Height scales and InBody 270 bioimpedance measurements will be used to assess body mass, lean mass, fat mass, fat percentage, and BMI z-score.

Muscular fitness and motor control. The horizontal countermovement jump test, arrowhead agility test, the stork balance test and the handgrip strength test will be used to assess muscular fitness and motor control.

To investigate the potential impact of the FIT FIRST Teen program on students' well-being and body perceptions, a series of questionnaires will be used.

Health-Related Quality of Life will be assessed using the KIDSCREEN-27. To investigate adolescents' body image, the Body Appreciation Scale will be employed. The Functionality Appreciation Scale will be used to measure such an outcome. The Perceived Locus of Causality Scale will be used to examine adolescents' motivational regulation towards physical education. Finally, the physical self-perception will be measured using the Physical Self-Inventory.

A mixed-method approach will be used to investigate the FIT FIRST Teen implementation, fidelity, acceptability, appropriateness, and feasibility. Questionnaires, semi-structured interviews, and logbooks will be employed by the research team.

ELIGIBILITY:
Inclusion Criteria:

* part of the enrolled classes

Exclusion Criteria:

* none

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 912 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiometabolic Fitness | Change from baseline to 40 weeks
  The cardiometabolic fitness profile will be evaluated by using the Yo-Yo test measured as the total distance in meters as an indicator for the participants' ability to perform intermittent exercise and their cardiometabolic fitness. The longer the distance, the better the cardiometabolic fitness of the participants.
Implementation | From baseline to 40 weeks
  Implementation of the FIT FIRST Teen Program will be evaluated.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Change from baseline to 40 weeks
  Health-Related Quality of Life will be measured using the KIDSCREEN-27 inventory.
Body Image | Change from baseline to 40 weeks
  Adolescents' body image will be measured using the Body Appreciation Scale-2.
Body Functionality Appreciation | Change from baseline to 40 weeks
  Adolescents' body functionality appreciation will be measured using the Functionality Appreciation Scale.
Motivation towards Physical Education | Change from baseline to 40 weeks
  Adolescents' motivational regulation towards physical education will be assessed using the Perceived Locus of Causality Scale.
Body Self-perception | Change from baseline to 40 weeks
  Adolescents' physical self-perception will be measured using the Physical Self-Inventory.
Resting Heart Rate | Change from baseline to 40 weeks
  Resting heart rate will be measured at rest. We will conduct 3 measurements after an 8-minute resting period
Blood Pressure | Change from baseline to 40 weeks
  Blood Pressure will be measured at rest. We will conduct 3 measurements after an 8-minute resting period
Muscular Fitness | Change from baseline to 40 weeks
  To investigate muscular fitness, the horizontal countermovement jump will be used to assess the lower body strength.
Muscular Fitness | Change from baseline to 40 weeks
  To investigate muscular fitness, the the handgrip test will be employed to evaluate the upper body strength.
Muscular Fitness | Change from baseline to 40 weeks
  To investigate muscular fitness, the Arrowhead agility test will be used.
Muscular Fitness | Change from baseline to 40 weeks
  To investigate postutal balance, the stork test will be used.
Body Composition | Change from baseline to 40 weeks
  InBody 270 bioimpedance will be used to measure body composition.
Height | Change from baseline to 40 weeks
  Tanita Height scales will be used to measure height.

CONTACTS AND LOCATIONS:
Locations (1):
- Rosengårdskolen, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided